CLINICAL TRIAL: NCT04130581
Title: Exercising the Motor Cortex Using Brain Stimulation
Brief Title: Brain Stimulation During Arm Immobilisation
Acronym: ImmobiStim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Helen Nuttall, Lecturer in Cognitive Neuroscience, Lancaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PSA1775
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Muscle Loss
MeSH Terms: conditions — Muscular Atrophy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS (Experimental): Six 30-pulse trains of 20 Hz repetitive Transcranial Magnetic Stimulation to left primary motor cortex hand area, separated by 60 seconds, repeated at 0, 24, 48, and 72 hours post-immobilisation.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)
- Sham (Sham Comparator): Six 30-pulse trains of 20 Hz repetitive sham Transcranial Magnetic Stimulation above, but not in contact with, the head, separated by 60 seconds, repeated at 0, 24, 48, and 72 hours post-immobilisation.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — TMS is a safe and non-invasive technique, which involves the generation of brief magnetic pulses applied to the head through a coil. The magnetic pulses pass through the scalp and skull and induce weak electric currents in the neural tissue directly underneath the coil. When TMS is applied in repetitive, patterned trains of pulses (rTMS), it can induce cortical plasticity specifically in the targeted brain region.

SUMMARY:
The research project explores how non-invasive brain stimulation can be used to detect and ameliorate loss of muscle strength after inactivity. At present, there is a limited understanding of how to maintain muscle strength during inactivity. Increasing evidence indicates that reduction in muscle strength following immobilisation is associated with reduced cortical motor output. Therefore, the aim of the study is to test if brain stimulation, can maintain cortical motor output and ameliorate the loss of muscle strength following immobilisation.

ELIGIBILITY:
Inclusion Criteria:

* Male
* right-handed
* aged 18-30
* healthy BMI

Exclusion Criteria:

* no primary muscle disorders
* no open wounds or skin conditions to arms and hands
* no neurological disorders or history of
* no history of fainting/convulsions
* no metal implanted into head/eye/neck
* non-smoker
* no arm, hand, fingers, shoulder injuries

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Motor Evoked Potentials (MEPs) across time points | 0, 24, 48, and 72 hours
  MEPs are elicited via TMS to primary motor cortex and index the excitability of the motor pathway. They are recorded non-invasively from muscles using surface electrodes. At each time point of the study (0, 24, 48, 72 hours) record MEPs will be recorded pre and post-intervention from the hand muscles of the dominant (immobilised) arm, and non-dominant (non-immobilised arm), to evaluate changes in excitability. Specifically, the peak-to-peak value of the MEPs from the hand will be measured, which reflects the amplitude of the MEP response. The latency of the MEP to index neural conduction speed will also be measured.

SECONDARY OUTCOMES:
Change in grip strength across time points | 0, and 72 hours.
  Grip strength of the dominant and non-dominant hands will be assessed using an isokinetic dynamometer at 0 and 72 hrs post-immobilisation. This will measure the strength of the hand muscles.

CONTACTS AND LOCATIONS:
Locations (1):
- Lancaster University, Lancaster, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No